CLINICAL TRIAL: NCT03471819
Title: Serotonin Levels in Atopic Dermatitis Patients and Its Relation to Disease Severity
Brief Title: Serotonin Levels in Atopic Dermatitis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Mohamed Abdelbary, Principal Investigator, Assiut University
Other Study IDs: SLAD
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Dermatologic Disease
Keywords: Atopic Dermatitis; serotonin
MeSH Terms: conditions — Skin Diseases; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients withf Atopic Dermatitis: Diagnosis is based upon American Academy of Dermatology recommendations for Diagnostic Criteria 2014.
  Interventions: Diagnostic Test: Serum serotonin level
- healthy volunteers: Normal individuals not complaining of any dermatological diseases
  Interventions: Diagnostic Test: Serum serotonin level

INTERVENTIONS:
Diagnostic Test: Serum serotonin level — blood sample will be obtained to evaluate serum level of serotonin

SUMMARY:
Atopic dermatitis (AD) is a chronic pruritic inflammatory skin disease of unknown aetiology. Global prevalence rates range from 1%-20%.AD is often worsened by stress and anxiety.Plasma levels of 5-HT were found to be positively correlated with the disease severity.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic pruritic inflammatory skin disease of unknown aetiology. The condition typically starts in infancy with changing presentations over the years. Incessant pruritus is the main symptom.

Main findings include: xerosis, eczematous lesions, Ig E reactivity, relapsing course and personal or family history of other atopic diatheses .Global prevalence rates range from 1%-20%.

AD is often worsened by stress and anxiety. Moreover, a mutual relationship between the neuroendocrine system and the immune system; including the skin has been suggested. Different mediators are responsible for this relation. Serotonin is considered as one of the most important responsible mediators (5-hydroxy-tryptamine; 5-HT) .

Patients with AD have been reported to have high serum levels of 5-HT. Moreover, plasma levels of 5-HT were found to be positively correlated with the disease severity. However and to the best of the investigators' knowledge, no studies have addressed this point in Egypt.

Treatment of AD includes: Elimination of triggers, emollients, topical therapies, and systemic modalities including SSRIs (Selective Serotonin Reuptake Inhibitors) and TCAs (Tricyclic Antidepressants) in certain cases. SSRIs block the reuptake of serotonin, thus increase the concentration of serotonin within synaptic clefts. The mechanism of action in relation to pruritus is not understood, but SSRIs have been used to treat atopic dermatitis associated pruritus

ELIGIBILITY:
Inclusion Criteria:

* All patients with the clinical diagnosis of AD.
* Age more than 2

Exclusion Criteria:

* Age less than 2 years.
* Any concomitant systemic or dermatological disease.
* Patients on any topical or systemic treatment during the past one month.
* Uncooperative patients.
* Refusal to participate

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 patients with the clinical diagnosis of AD and 30 age and sex-matched apparently healthy volunteers will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
SCORAD | one month
  Scoring Atopic Dermatitis "SCORAD" is a clinical tool for assessing the severity of AD as objectively as possible.
  It includes:
  A: Spread B: Intensity C: Subjective symptoms

SECONDARY OUTCOMES:
Beck's depression score (Arabic version) | one month
  its a psychiatric 13 items questionnaire to determine the severity of depression

CONTACTS AND LOCATIONS:
Overall Officials: Dalia A Negm, Lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdel-Hafez K, Abdel-Aty MA, Hofny ER. Prevalence of skin diseases in rural areas of Assiut Governorate, Upper Egypt. Int J Dermatol. 2003 Nov;42(11):887-92. doi: 10.1046/j.1365-4362.2003.01936.x. PMID 14636205
- [Background] Gooderham MJ, Hong HC, Eshtiaghi P, Papp KA. Dupilumab: A review of its use in the treatment of atopic dermatitis. J Am Acad Dermatol. 2018 Mar;78(3 Suppl 1):S28-S36. doi: 10.1016/j.jaad.2017.12.022. PMID 29471919
- [Background] Afzal R, Shim WS. Glucosylsphingosine Activates Serotonin Receptor 2a and 2b: Implication of a Novel Itch Signaling Pathway. Biomol Ther (Seoul). 2017 Sep 1;25(5):497-503. doi: 10.4062/biomolther.2016.207. PMID 28208011